CLINICAL TRIAL: NCT05832892
Title: A Phase Ib/II Clinical Trial to Evaluate the Efficacy and Safety of Surufatinib in Combination With KN046 and AG Regimen Chemotherapy for the First-Line Treatment of Unresectable Advanced Pancreatic Cancer
Brief Title: Surufatinib Combined With KN046 and AG Regimen Chemotherapy as First-Line Treatment for Unresectable Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSPAC-02
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-06

CONDITIONS: Unresectable Locally Advanced or Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer; Surufatinib; KN046; Nab-paclitaxel; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — surufatinib; Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- surufatinib + KN046 + nab-paclitaxel + gemcitabine (Experimental): In the phase Ib of dose escalation, all patients enrolled will receive: nab-paclitaxel at 125 mg/m2 on days 1 and 8, gemcitabine at 1000 mg/m2 on days 1 and 8, KN046 at 5 mg /kg on day 1, plus surufatinib per cohort escalation assignment starting with 200 mg. The combination treatment repeats every 3 weeks, until disease progression, death, intolerable toxicity, or withdrawal of informed consent. Dose-limiting toxicity will be evaluated 28 days after first dose to determine the recommended phase 2 dose (RP2D) of surufatinib.
  Patients enrolled in the phase II of dose expansion will receive the combination regimen of nab-paclitaxel plus gemcitabine plus KN046 plus surufatinib as determined in the phase Ib.
  Interventions: Drug: surufatinib; Drug: KN046; Drug: gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: surufatinib — In phase Ib, surufatinib will be orally administrated 200 mg once a day (QD) or 250 mg QD per cohort escalation assignment on a 21-day cycle.
  In phase II, surufatinib will be orally administrated at RP2D as determined in phase Ib.
  Other Names: HMPL-012; Sulfatinib
Drug: KN046 — Nab-paclitaxel will be administrated at 125 mg/m2 intravenously on day 1 and 8 of each 21-day cycle.
Drug: gemcitabine — Gemcitabine will be administrated at 1000 mg/m2 intravenously on day 1 and 8 of each 21-day cycle.
  Other Names: GEMZAR
Drug: Nab paclitaxel — Nab-paclitaxel will be administrated at 125 mg/m2 intravenously on day 1 and 8 of each 21-day cycle.
  Other Names: nanoparticle albumin-bound paclitaxel; Abraxane; ABI-007

SUMMARY:
Advanced pancreatic cancer is a highly aggressive and fatal disease with an extremely low 5-year survival rate. Combined chemotherapy is the mainstay of treatment for patients with unresectable advanced pancreatic cancer, and the combination of nab-paclitaxel and gemcitabine (AG regimen) has been one of the most commonly used regimens for more than a decade. However, chemo-resistance often occurs within half a year and the efficacy remains unsatisfied with an overall survival of only 9~11 months.

Immune checkpoint inhibitors (ICIs) such as anti-PD-1/L1 antibody and anti-CTLA-4 antibody have demonstrated encouraging anti-tumor efficacy in multiple solid tumors including lung cancer, gastric cancer, and esophageal cancer, while obtained controversial results when combined with chemotherapy in pancreatic cancer. Recently, the immune-suppression tumor microenvironment (TME) of pancreatic cancer has been described in several pre-clinical studies, which may explain the resistance against ICIs and chemotherapy.

KN046 is a recombinant humanized PD-L1/CTLA-4 bispecific antibody with innovative designs include a proprietary CTLA-4 domain antibody with a significantly improved safety profile, a bispecific antibody fused with PD-L1 antibody targeting the TME with high PD-L1 expression. Recent clinical studies have shown promising anti-tumor activity of KN046 in pancreatic cancer.

Surufatinib, also known as HMPL-012 or Sulfatinib, is a small molecular tyrosine kinase inhibitor (TKI) targeting the Vascular Endothelial Growth Factor Receptor (VEGFR), Fibroblast Growth Factor Receptor (FGFR) and Colony Stimulating Factor-1 Receptor (CSF-1R), which has a dual mechanism of action of anti-angiogenesis and regulation of immune microenvironment. Previous studies have suggested synergic effect of surufatinib in combination with anti-PD-1 antibodies.

This phase Ib/II clinical trial is intended to investigate the activity and safety of the combination of surufatinib combined with KN046 and the AG regimen chemotherapy as first-line treatment in patients with unresectable locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Advanced pancreatic cancer is a highly aggressive and fatal disease with an extremely low 5-year survival rate. Combined chemotherapy is the mainstay of treatment for patients with unresectable advanced pancreatic cancer, and the combination of nab-paclitaxel and gemcitabine (AG regimen) has been one of the most commonly used regimens for more than a decade. However, chemo-resistance often occurs within half a year and the efficacy remains unsatisfied with an overall survival of only 9~11 months.

Immune checkpoint inhibitors (ICIs) such as anti-PD-1/L1 antibody and anti-CTLA-4 antibody have demonstrated encouraging anti-tumor efficacy in multiple solid tumors including lung cancer, gastric cancer, and esophageal cancer, while obtained controversial results when combined with chemotherapy in pancreatic cancer. Recently, the immune-suppression tumor microenvironment (TME) of pancreatic cancer has been described in several pre-clinical studies, which may explain the resistance against ICIs and chemotherapy.

KN046 is a recombinant humanized PD-L1/CTLA-4 bispecific antibody with innovative designs include a proprietary CTLA-4 domain antibody with a significantly improved safety profile, a bispecific antibody fused with PD-L1 antibody targeting the TME with high PD-L1 expression. Recent clinical studies have shown promising anti-tumor activity of KN046 in pancreatic cancer.

Surufatinib, also known as HMPL-012 or Sulfatinib, is a small molecular tyrosine kinase inhibitor (TKI) targeting the Vascular Endothelial Growth Factor Receptor (VEGFR), Fibroblast Growth Factor Receptor (FGFR) and Colony Stimulating Factor-1 Receptor (CSF-1R), which has a dual mechanism of action of anti-angiogenesis and regulation of immune microenvironment. Previous studies have suggested synergic effect of surufatinib in combination with anti-PD-1 antibodies.

This phase Ib/II clinical trial is intended to investigate the activity and safety of the combination of surufatinib combined with KN046 and the AG regimen chemotherapy as first-line treatment in patients with unresectable locally advanced or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment.
* Male or female, age ≥ 18 years and ≤ 75 years.
* Patients must have histologically or cytologically confirmed pancreatic adenocarcinoma that originated from the pancreatic ductal epithelial, with image-documented unresectable locally advanced or distant metastatic disease.
* Patients have received no previous local treatment such as surgery, radiotherapy, ablation, or any systemic treatment for advanced/metastatic pancreatic cancer, including neoadjuvant and/or adjuvant therapy.
* Have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected overall survival of ≥ 6 months.
* Laboratory test results within 7 days prior to first dose of study drugs must meet the following criteria:

  1. absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L and hemoglobin (HGB) ≥ 90 g/L.
  2. total bilirubin (TBil) ≤ 1.5 × the upper limit of normal (ULN).
  3. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN in the absence of liver metastases; ALT and AST ≤ 3 × ULN in the presence of liver metastases.
  4. serum creatinine (SCr) ≤ 1.5 × ULN and creatinine clearance (CCl) ≥ 50 mL/min (calculated according to the Cockcroft-Gault formula).
  5. urine protein <2+ in urine analysis; if urine protein ≥2+, 24-hour urine protein quantification should be <1g.
  6. international normalized ratio (INR) ≤ 1.5 and partial activation prothrombin time (APTT) ≤ 1.5 × ULN.
* Female subjects of childbearing age or male subjects whose partner is a female of childbearing age should use effective contraception from at least 1 month prior to the first dose of study drugs to 6 months after the last dose of study drugs.

Exclusion Criteria:

* Adverse events (AEs) due to previous anti-tumor therapy have not recovered to CTCAE Grade ≤1 (except for hair loss, skin pigment changes, or Grade ≤ 2 neurotoxicity).
* Other malignancies diagnosed within past 5 years (except basal cell carcinoma of the skin or squamous cell carcinoma and carcinoma in situ of the cervix that have been effectively controlled).
* Presence of central nervous system (CNS) metastases at screening, or have a history of CNS metastases.
* Patients who have received approved systemic anti-tumor therapy within 4 weeks before the first dose of study drugs, including chemotherapy, biological therapy, targeted therapy, hormone therapy, traditional Chinese medicine therapy (with clear anti-tumor indications in the label), etc.
* Patients who have received radical radiotherapy (including radiotherapy involving > 25% bone marrow) within 4 weeks prior to the first study drugs reception; Or brachytherapy (e.g., implanted radioparticles) within 60 days prior to the first dose of the study drugs; Or palliative radiotherapy for bone metastases within 1 week prior to first dose of the study drugs.
* Patients who have undergone major surgery within 4 weeks before receiving first dose of study drugs, or have unhealed wounds, ulcers or fractures.
* Vaccination within 4 weeks before the first dose of study drugs or plan to have during the study period, except for inactivated vaccines.
* Patients who have previously received anti-VEGF/VEGFR agents and have experienced disease progression during treatment or within 3 months after the last dose.
* Patients with uncontrollable malignant pleural effusion, ascites, or pericardial effusion (no response to diuretics or puncture as per the investigator's judgement).
* Presence of gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding in unresected tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by the investigator.
* Patients with evidence or history of thrombosis or significant bleeding tendency (bleeding >30 mL within 2 months, hematemesis, melena, hematochezia, or hemoptysis >5mL within 4 weeks) within 2 months prior to the first dose of the study drugs.
* Patients who have arterial thrombosis or deep vein thrombosis within 6 months, or have thromboembolic events (including stroke and/or transient ischaemic attack) within 12 months prior to first dose of the study drugs.
* Patients who are receiving anti-tuberculosis therapy for active pulmonary tuberculosis, or have had anti-tuberculosis therapy within 1 year prior to first dose of the study drugs.
* Patients with a previous or current history of pulmonary disorder that may interfere the identification and management of suspected drug-related pulmonary toxicity, including pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc. (radiation pneumonia in radiotherapy areas is allowed).
* Presence of corneal lesions, including but not limited to bullous keratopathy, shingle corneal degeneration, corneal abrasions, corneal ulcers, keratitis, etc.
* History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive; known Hepatitis C virus (HCV) infection with HCV RNA positive; or other hepatitis, liver cirrhosis, etc.
* Positive for human immunodeficiency virus (HIV) antibodies.
* Meet any of the following criteria for cardiac function:

  1. Clinically significant arrhythmias or conduction abnormalities requiring clinical intervention.
  2. Electrocardiogram (ECG) indicating an QT interval (QTcF) of > 480 msec.
  3. Clinically significant cardiovascular diseases, including acute myocardial infarction within 6 months prior to enrollment, severe/unstable angina pectoris, coronary artery bypass grafting, congestive heart failure according to the New York Heart Association (NYHA) classification III/IV, ventricular arrhythmias needing drug intervention, LVEF <50%.
* Previous or current autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener syndrome, Graves' disease, rheumatoid arthritis, pituitary inflammation, ocular pigmentitis, autoimmune hepatitis, systemic sclerosis, Hashimoto's thyroiditis, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome), with exceptions as follows: type I diabetes, hormone replacement therapy-stabilized hypothyroidism, psoriasis or vitiligo that does not require systemic therapy.
* Women who are pregnant or lactating.
* Known history of allergy to the relevant ingredients of the study drugs.
* Subjects who have received investigational treatments in other clinical studies within 4 weeks prior to first dose of study drugs.
* Patients who have any disorder or condition that may affect absorption of the study drugs, or who are unable to take oral medication.
* Patients unsuitable for participating due to other reasons as per investigator's determination.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (RECIST 1.1) | From date of first dose until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 24 months
  ORR is defined as the percentage of patients who achieve complete response (CR) or partial response (PR) based on the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Objective response rate (irRECIST) | From date of first dose until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 24 months
  It will be evaluated based on the immune-related (ir) RECIST criteria.
Disease control rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 24 months
  DCR is defined as the percentage of patients who achieved CR, PR and stable disease (SD), and will be evaluated based on RECIST 1.1 and the irRECIST criteria.
Duration of response (RECIST 1.1) | From date of first dose until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 24 months
  DoR is defined as the time from first documented objective response (CR or PR, whichever occurs first, as per RECIST v1.1) to disease progression or death, whichever occurs first.
Progression free survival (RECIST 1.1) | From date of first dose until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 24 months
  PFS is defined as the time from the date of first dose of study drugs to the date of the first documented disease progression (determined as per RECIST v1.1) or date of death, whichever occurs first.
Overall survival | From date of first dose until the date of death from any cause, assessed up to 24 months
Safety and tolerability by incidence, severity and outcome of adverse events | From first dose to within 90 days after the last dose, up to 24 months
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTCAE Version 5.0.
  Dose-limiting toxicities (DLT) will be evaluated by the investigators 28 days after the first dose of study drugs in order to determine the RP2D of surufatinib in combination with KN046 and the AG regimen in phase Ib.
Predictive biomarkers | From date of screening until the date of death, assessed up to 24 months
  To evaluate the correlation between potential biomarkers and the prognosis of patients treated with this regimen. Tumor tissue or blood samples will be examined to assess relevant parameters including MSI/dMMR status, TMB, PD-1/PD-L1/CTLA-4 expression, VEGFR/FGFR/CSF-1R expression, plasma ctDNA, tumor markers such as CA19-9/CEA before and after treatment, plasma concentration of sVEGFR2, VEGF, FGF23, FGF2, M-CSF, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers in order to protect patients' privacy.